CLINICAL TRIAL: NCT05002868
Title: A Multi-center, Open-label, Phase I/Ib Study to Assess the Safety, Pharmacokinetics and Anti-tumor Activity of RP12146, a Poly (ADP-ribose) Polymerase (PARP) Inhibitor, in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Safety, Pharmacokinetics and Anti-tumor Activity of RP12146, in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP12146-2101
Record Dates: First submitted 2021-08-05; First posted 2021-08-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor; Extensive-stage Small-cell Lung Cancer; Locally Advanced Breast Cancer; Metastatic Breast Cancer; Platinum-sensitive Ovarian Cancer; Platinum-Sensitive Fallopian Tube Carcinoma; Platinum-Sensitive Peritoneal Cancer
Keywords: PARP
MeSH Terms: conditions — Small Cell Lung Carcinoma; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RP12146 (Experimental): RP12146 will be administered orally daily (QD or BID)
  Interventions: Drug: RP12146

INTERVENTIONS:
Drug: RP12146 — starting dose of 100 mg QD

SUMMARY:
An open-label, two-part Phase I/Ib study of RP12146 in adult patients with locally advanced or metastatic solid tumors. The first part (Part 1) is a Phase I dose-escalation, 3+3 design, open-label, MTD determination study and will enroll patients who have tumors known to harbour DNA repair deficiencies. The second part (Part 2) is a Phase Ib, dose-expansion at the MTD (or optimal dose) and will enroll patients with a confirmed deleterious HRR mutation in their tumor as identified by a central genomics testing laboratory.

ELIGIBILITY:
Inclusion Criteria.

1. Provision of full informed consent prior to any study-specific procedures.
2. Patients must be ≥18 years of age, at the time of signing informed consent.
3. Dose escalation phase, patients with histologically and/or cytologically confirmed malignant solid tumor whose disease has progressed following at least one standard therapy and who have no other acceptable standard treatment options. Tumor types will include breast, ovarian, fallopian tube, or peritoneal cancer, extensive-stage small cell lung cancer (ES-SCLC), prostate, pancreatic, colorectal gastric, biliary tract, and endometrial cancer.
4. Dose-expansion phase patients with histologically and/or cytologically confirmed malignant solid tumor (breast, ovarian, fallopian tube, or peritoneal cancer, extensive-stage small cell lung cancer (ES-SCLC), with one of the documented deleterious mutations of specified HRR genes and whose disease has progressed following at least one standard therapy.
5. Patients with at least one measurable lesion per RECIST version 1.1 at baseline that can be accurately assessed by CT-scan or MRI and is suitable for repeated assessment at follow up-visits.
6. ECOG performance status 0 to 2.
7. Use of contraception measures

Exclusion Criteria:

1. Patients with HER2 positive breast cancer
2. Patients receiving anticancer therapy
3. Patient who has not recovered from acute toxicities of previous therapy except treatment-related alopecia.
4. Prior treatment with a PARP inhibitor
5. Major surgery within 4 weeks of starting study treatment or any patient who has not recovered from the effects of major surgery.
6. Patient with symptomatic uncontrolled brain metastasis.
7. Pregnancy and lactation
8. Patients with uncontrolled disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of RP12146 in patients with locally advanced or metastatic solid tumors | 28 days
  The MTD was defined as the highest dose level at which no more than 1 in 6 participants experienced a dose-limiting toxicity (DLT) during the first 28-day cycle of treatment
Number of Participants With Treatment-emergent Adverse Events as Assessed by CTCAE Criteria v5.0 | 2 years
  Summary of Treatment-Emergent Adverse Events-(Causality All). Patients will be monitored for adverse events and both related and as well as non-related adverse events will be captured during the study. All adverse events (irrespective of causality) will be reported.

SECONDARY OUTCOMES:
Tmax | Day 1 to Day 28
  Pharmacokinetics: Time to Reach Maximum Concentration (Tmax) of RP12146
Cmax | Day 1 to Day 28
  Pharmacokinetics: Maximum Concentration (Cmax) of RP12146
AUC | Day 1 to Day 28
  Pharmacokinetics: Area Under the Concentration Curve (AUC) of RP12146
Overall response rate (ORR) | 2 years
  Sum of the percentages of Complete Response and Partial Response
Clinical benefit rate (CBR) | 2 years
  Sum of the percentages of Complete response, partial response and stable disease
Progression free survival (PFS) | 2 years
  It is defined as time from the first dose of study treatment to documented disease progression

CONTACTS AND LOCATIONS:
Locations (6):
- Multiscan s.r.o., Hořovice, Czechia
- Poland (5):
  - SP ZOZ University Hospital in Krakow Oncology Clinic, 50 Kopernika Street, Krakow
  - Klinika Onkologii ICZMP, Lodz
  - Pratia Poznań Medical Center, Poznan
  - Clinical Trials Site Nasz Lekarz, Torun
  - Maria Skłodowska-Curie Memorial National Oncology Institute, Warsaw

IPD SHARING:
Plan to Share IPD: No